CLINICAL TRIAL: NCT01620658
Title: Radioprotective Light-weight Caps in the Interventional Cardiology Setting: a Randomized Controlled Trial
Brief Title: Radioprotective Light-weight Caps in the Interventional Cardiology Setting
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Principal Investigator, Raul Herrera, MD, Director, Division of Clinical Research & Outcomes, Baptist Health South Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PROTECT
Record Dates: First submitted 2012-06-06; First posted 2012-06-15 (Estimated); Results first posted 2021-10-21 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-09

CONDITIONS: Occupational Exposure to Radiation
Keywords: Occupational Exposure to Radiation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard cap (Active Comparator): Interventionalist wear a standard fabric cap during fluoroscopy guided interventions.
  Interventions: Device: Standard cap
- 0.3mm XPF cap (Experimental): Interventionalist wear a XPF 0.3mm lead equivalent cap during fluoroscopy guided interventions.
  Interventions: Device: 0.3mm XPF cap
- 0.5mm XPF cap (Experimental): Interventionalist wear a XPF 0.5mm lead equivalent cap during fluoroscopy guided interventions.
  Interventions: Device: 0.5mm XPF cap

INTERVENTIONS:
Device: 0.5mm XPF cap — Interventionalist wear a XPF 0.5mm lead equivalent cap during fluoroscopy guided interventions.
  XPF is a trademark of BloXR (Salt lake City, UT) for a new bi-layer (Barium/Bismuth) radiation attenuation material.
  Arms: 0.5mm XPF cap
Device: 0.3mm XPF cap — Interventionalist wear a XPF 0.3mm lead equivalent cap during fluoroscopy guided interventions.
  XPF is a trademark of BloXR (Salt lake City, UT) for a new bi-layer (Barium/Bismuth) radiation attenuation material.
  Arms: 0.3mm XPF cap
Device: Standard cap — Interventionalist wear a standard fabric cap during fluoroscopy guided interventions.
  Arms: standard cap

SUMMARY:
The primary objective of the present trial is to compare the radiation attenuation provided by XPF caps (0.5mm lead-equivalent and 0.3mm lead-equivalent) to the standard protection (fabric cap, basically no protection) as measured in % radiation attenuation) during 150 days of fluoroscopy guided cardiology interventions. The second objective is to compare the operator comfort (rated on a visual analog scale) of wearing the XPF protection caps compared to the standard fabric caps.

DETAILED DESCRIPTION:
The primary objective of the present trial is to compare the radiation attenuation provided by XPF caps (0.5mm lead-equivalent and 0.3mm lead-equivalent) to the standard protection (fabric cap, basically no protection) as measured in % radiation attenuation) during 150 days of fluoroscopy guided cardiology interventions. The second objective is to compare the operator comfort (rated on a visual analog scale) of wearing the XPF protection caps compared to the standard fabric caps.

For more information please contact Dr. Raul Herrera, MD, Director Baptist Cardiac and Vascular Institute Baptist Hospital of Miami.

ELIGIBILITY:
Inclusion Criteria:

* Interventional Cardiologist practicing in Baptist Cardiac & Vascular Institute
* cardiac procedure requiring C-arm fluoroscopy

Exclusion Criteria:

* Interventional Neuroradiologists and Interventional Radiologists will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Herrera, MD, Principal Investigator — Baptist Hospital of Miami, Miami Cardiac and Vascular Institute
Locations (1):
- Baptist Hospital of Miami, Miami Cardiac and Vascular Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uthoff H, Quesada R, Roberts JS, Baumann F, Schernthaner M, Zaremski L, Hajirawala L, Katzen BT, Staub D, Kreusch AS. Radioprotective lightweight caps in the interventional cardiology setting: a randomised controlled trial (PROTECT). EuroIntervention. 2015 May;11(1):53-9. doi: 10.4244/EIJV11I1A9. PMID 25982649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to the Miami Cardiac and Vascular Institute for Imaging Study/Procedure.
Pre-assignment Details: Voluntary patient participation. PI responsible for patient selection.
Groups:
- 0.3mm XPF Cap: Interventionalist wear a XPF 0.3mm lead equivalent cap during fluoroscopy guided interventions.
  0.3mm XPF cap: Interventionalist wear a XPF 0.3mm lead equivalent cap during fluoroscopy guided interventions.
  XPF is a trademark of BloXR (Salt lake City, UT) for a new bi-layer (Barium/Bismuth) radiation attenuation material.
- 0.5mm XPF Cap: Interventionalist wear a XPF 0.5mm lead equivalent cap during fluoroscopy guided interventions.
  0.5mm XPF cap: Interventionalist wear a XPF 0.5mm lead equivalent cap during fluoroscopy guided interventions.
  XPF is a trademark of BloXR (Salt lake City, UT) for a new bi-layer (Barium/Bismuth) radiation attenuation material.
Period: Overall Study
Arm/Group | Standard Cap | 0.3mm XPF Cap | 0.5mm XPF Cap
Started | 59 | 74 | 64
Completed | 35 | 45 | 44
Not Completed | 24 | 29 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Cap | 0.3mm XPF Cap | 0.5mm XPF Cap | Total
Number analyzed (Participants) | 59 | 74 | 64 | 197
Age, Continuous [Mean (Full Range); unit: years] | 53 [40 to 65] | 53 [40 to 65] | 53 [40 to 65] | 53 [40 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 30 | 95
  Male | 30 | 38 | 34 | 102
Region of Enrollment [Number; unit: participants]
  United States | 59 | 74 | 64 | 197

OUTCOME MEASURES:

1. Primary Outcome: Radiation Attenuation in Percentage (%)
Description: The null hypothesis is that the XPF 0.5mm lead-equivalent caps attenuation is equal to the XPF 0.3mm lead-equivalent and standard cap attenuations. The alternative hypothesis is that the XPF 0.5mm lead-equivalent cap attenuation is superior or inferior to the XPF 0.3mm lead-equivalent and standard cap attenuations. The groups will be compared separately and a pooled analysis, comparing XPF 0.5mm and 0.3mm combined vs. standard is also planned.The radiation protection (radiation dose reduction) expressed as a percentage was calculated by subtracting radiation measured underneath the cap from radiation measured outside the cap and then dividing this difference by the product of radiation measured outside the cap multiplied by 100.
Time Frame: 1 day
Population: Mean Radiation Protection is described under Outcome Measure Data below.
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Standard Cap | 0.3mm XPF Cap | 0.5mm XPF Cap
Number analyzed (Participants) | 35 | 45 | 44
Percentage | 12 [4.9 to 19.1] | 91.5 [87.4 to 95.6] | 97.1 [92.5 to 100]

2. Primary Outcome: Absolute Radiation Exposure Outside of Cap
Description: The cumulative radiation doses were defined as the summation of all correspondent equivalent doses measured.
Time Frame: 1 day
Population: The primary objective of the trial is to show how much radiation attenuation is provided by XPF in absolute and relative terms.
Measure: Mean (95% Confidence Interval); unit: uSv
Groups:
- Radiation Exposure Monitored With Standard Caps.: Operators were randomly assigned to wear standard fabric Caps. Radiation doses were measured by using dosimeters placed outside and underneath the caps.
- Radiation Exposure Monitored With XPF 0.3 mm Caps: Operators were randomly assigned to wear the 0.3 mm Caps. Radiation doses were measured by using dosimeters placed outside and underneath the caps.
- Radiation Exposure Monitored With XPF 0.5mm Caps: Operators were randomly assigned to wear lead-equivalent XPF caps. Radiation doses were measured by using dosimeters placed outside and underneath the caps.
Arm/Group | Radiation Exposure Monitored With Standard Caps. | Radiation Exposure Monitored With XPF 0.3 mm Caps | Radiation Exposure Monitored With XPF 0.5mm Caps
Number analyzed (Participants) | 35 | 45 | 44
uSv | 132 [21 to 243] | 118 [54 to 183] | 59 [33 to 85]

3. Secondary Outcome: Operator Comfort Assessment
Description: After completion of the last procedure on each day, the operators were asked to rate the comfort of wearing the cap on a scale from 0 (unbearably heavy, badly fitting) to 100 (very light, well fitting).
Time Frame: 1 day per participant, a total of 197 operator days
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Standard Caps: Operators were randomly assigned to wear standard fabric Caps. The operator comfort rating on the VAS (score range, 0-100), with higher numbers indicating better comfort, was obtained in all cases and for all operators.
- XPF 0.3 mm: Operators were randomly assigned to wear XPF 0.3mm Caps. The operator comfort rating on the VAS (score range, 0-100), with higher numbers indicating better comfort, was obtained in all cases and for all operators.
- XPF 0.5 mm: Operators were randomly assigned to wear XPF 0.5mm Caps. The operator comfort rating on the VAS (score range, 0-100), with higher numbers indicating better comfort, was obtained in all cases and for all operators.
Arm/Group | Standard Caps | XPF 0.3 mm | XPF 0.5 mm
Number analyzed (Participants) | 59 | 74 | 64
score on a scale | 90 [0 to 100] | 90 [0 to 100] | 90 [0 to 100]

4. Secondary Outcome: Operator Comfort Assessment Based on Weight
Description: After completion of the last procedure on each day, the caps worn by the operators were weighed to assess comfort of wearing the standard cap, XPF 0.3mm and XPF 0.5mm caps. The operators were asked to rate the comfort of wearing the cap on a scale from 0 (unbearably heavy, badly fitting) to 100 (very light, well fitting).
Time Frame: 1 day per participant, a total of 197 operator days
Measure: Mean (Full Range); unit: grams
Arm/Group | Standard Caps | XPF 0.5 mm | XPF 0.3 mm
Number analyzed (Participants) | 59 | 64 | 74
grams | 12.5 [12.5 to 12.6] | 123.7 [122.9 to 124.6] | 118.4 [116.7 to 120.3]

ADVERSE EVENTS:
Arm/Group | Standard Cap | 0.3mm XPF Cap | 0.5mm XPF Cap
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/74 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/74 | 0/64
Other Adverse Events (participants affected / at risk) | 0/59 | 0/74 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No